CLINICAL TRIAL: NCT03586232
Title: Effects of Arnica Montana and Bromelain in Rhinoplasty
Brief Title: Arnica Montana and Bromelain in Rhinoplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be conducted since funding was not obtained.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-37291
Record Dates: First submitted 2018-07-03; First posted 2018-07-13 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Wound Healing
Keywords: Rhinoplasty; Arnica Montana; Bromelain; Body healing post op; Rhinoplasty Outcome Evaluation
MeSH Terms: interventions — Arnicae flos extract; Bromelains

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Participants will take two placebo pills q8 hours for 7 days preoperatively and 7 days postoperatively, in addition to the standard postoperative tapered methylprednisolone.
  Interventions: Other: Placebo
- Arnica Montana (Experimental): Participants will take Arnica Montana, 30C oral, pill and a placebo pill q8 hours for 7 days preoperatively and 7 days postoperatively, in addition to the standard postoperative tapered methylprednisolone.
  Interventions: Dietary Supplement: Arnica Montana; Other: Placebo
- Arnica Montana and Bromelain (Experimental): Participants will take Bromelain, 500mg oral pill + Arnica Montana, 30C oral, q8 hours for 7 days preoperatively and 7 days postoperatively, in addition to the standard postoperative tapered methylprednisolone.
  Interventions: Dietary Supplement: Arnica Montana; Dietary Supplement: Bromelain

INTERVENTIONS:
Dietary Supplement: Arnica Montana — Arnica Montana is from the Asteraceae plant family and is native to the mountain areas in Europe and western North America. It is reported to have anti-inflammatory, antiseptic, and vasodilatory properties and is often used in plastic surgery to help reduce pain, edema, and ecchymosis postoperatively.
  Arms: Arnica Montana; Arnica Montana and Bromelain
Dietary Supplement: Bromelain — Bromelain is a protease enzyme derived from the pineapple plant, Ananas comosus, which has been used to reduce swelling, inflammation, and pain and may help to reduce wound healing time.
  Arms: Arnica Montana and Bromelain
Other: Placebo — A pharmacologically inert preparation
  Arms: Arnica Montana; Control

SUMMARY:
The purpose of this study is to assess the perioperative use of Arnica Montana and the combined use of Arnica Montana and Bromelain in aiding the body's wound healing functions during the postoperative period after rhinoplasty. The secondary objective of the study is to determine if there is a reduction in postoperative edema when Arnica Montana and Bromelain are combined. Another secondary objective is to demonstrate increased patient satisfaction with the use of Arnica Montana and the combination Arnica Montana and Bromelain.

ELIGIBILITY:
Inclusion Criteria:

-adults scheduled for outpatient primary rhinoplasty with osteotomies at Boston Medical Center

Exclusion Criteria:

* oral or contact allergies to Arnica Montana or to derivatives from the Ananas comosus or to any other member of the Asteraceae family of plants such as ragweed, chrysanthemums, marigolds, and daisies or Bromelain as determined by self disclosure.
* allergies to pineapple as Bromelain is from pineapple extract
* currently taking antiplatelet medication or anticoagulation medications
* chronic use of NSAIDs meaning those currently using NSAIDS daily for at least 3 months
* taking other homeopathic remedies during the perioperative period
* bleeding disorders as determined by self-disclosure or strong family history, patients in question who would like to participate in the study will have blood work obtained prior to operation
* chronic medical conditions such as significant pulmonary, cardiac, liver, or kidney disease are excluded including poorly controlled hypertension or patients on more than one antihypertensive agent and patients with diabetes
* malignancy, infection, immunodeficiency, metabolic syndrome, infectious, or inflammatory gastrointestinal disease
* severe liver or kidney disease
* significant psychiatric disorders
* females who are breast feeding or pregnant
* history of nasal surgery
* history of head and neck malignancy
* taking oral corticosteroid therapy
* undergoing additional surgery other than primary rhinoplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Ecchymosis extent 7 days post rhinoplasty | 7 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the ecchymosis from 0-5 where 0= no ecchymosis, 1= up to medial one third of the lower and or upper eyelid, 2=medial half of the upper and or lower eyelid, 3=entire upper and lower eyelid, 4= entire lower and upper eyelid and or conjunctive, 5= extension of ecchymosis below the molar bone. Lower scores are more favorable.
Ecchymosis extent 14 days post rhinoplasty | 14 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the ecchymosis from 0-5 where 0= no ecchymosis, 1= up to medial one third of the lower and or upper eyelid, 2=medial half of the upper and or lower eyelid, 3=entire upper and lower eyelid, 4= entire lower and upper eyelid and or conjunctive, 5= extension of ecchymosis below the molar bone. Lower scores are more favorable.
Ecchymosis extent 28 days post rhinoplasty | 28 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the ecchymosis from 0-5 where 0= no ecchymosis, 1= up to medial one third of the lower and or upper eyelid, 2=medial half of the upper and or lower eyelid, 3=entire upper and lower eyelid, 4= entire lower and upper eyelid and or conjunctive, 5= extension of ecchymosis below the molar bone. Lower scores are more favorable.
Ecchymosis color density 7 days post rhinoplasty | 7 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the the color density (intensity) of the ecchymosis from 0-5 where 0=no color change, 1= yellowish color change, 3: light purple, 4: dark purple, 5: very dark purple.Lower scores are more favorable.
Ecchymosis color density 14 days post rhinoplasty | 14 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the the color density (intensity) of the ecchymosis from 0-5 where 0=no color change, 1= yellowish color change, 3: light purple, 4: dark purple, 5: very dark purple.Lower scores are more favorable.
Ecchymosis color density 28 days post rhinoplasty | 28 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the the color density (intensity) of the ecchymosis from 0-5 where 0=no color change, 1= yellowish color change, 3: light purple, 4: dark purple, 5: very dark purple.Lower scores are more favorable.
Edema 7 days post rhinoplasty | 7 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1 frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the edema from 0-3 where 0=no edema, 1=mild edema, 2= moderate edema 3= severe edema. Lower scores are more favorable.
Edema 14 days post rhinoplasty | 14 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1 frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the edema from 0-3 where 0=no edema, 1=mild edema, 2= moderate edema 3= severe edema. Lower scores are more favorable.
Edema 28 days post rhinoplasty | 28 days
  Blinded facial plastic surgeons will review 4 photographs of participants (1 frontal, 2 oblique, and 1 nasal base view) and using the photo analysis scale by Totonchi and Guyuron assign each participant an average score based on the extent of the edema from 0-3 where 0=no edema, 1=mild edema, 2= moderate edema 3= severe edema. Lower scores are more favorable.

SECONDARY OUTCOMES:
Change in patient satisfaction | baseline, 28 days
  Participants will complete the validated Rhinoplasty Outcome Evaluation (ROE) at their initial consultation visit (preoperative responses) which will be compared to their postoperative survey to assess overall patient satisfaction in regards to their rhinoplasty one month postoperatively. The ROE questionnaire has 6 questions, each with 5 answer options, graded from 0 to 4 so scores can range from 0 to 24. In order to make understanding easier, the score obtained must be divided by 24 and multiplied by 100, which leads to a score varying between zero and 100, and the higher the score, the greater is the patient's satisfaction with the nose surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Wulu, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No